CLINICAL TRIAL: NCT02270684
Title: Comparative Effectiveness of an Activity-Specific Monitoring Device (StepRite) on Short Term Outcomes in Adults After Total Knee Arthroplasty
Brief Title: StepRite Evaluation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and retention difficulties
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Christopher Powers, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FP00002312; HS-13-00319 (Other: USC IRB)
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis
Keywords: Total Knee Arthroplasty; Home monitoring
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device (Experimental): Participants in this arm will receive the StepRite device. They will have a remote visit with their Physical Therapist in place of one in-person visit per week during the outpatient phase of their treatment
  Interventions: Device: StepRite
- Usual and customary care (No Intervention): Participants in this arm will undergo usual care and will not be issued with the StepRite device

INTERVENTIONS:
Device: StepRite — The StepRite device uses an insole to monitor motion, and relays this information to the physical therapist via a smart phone app and web link. Set exercises can be programmed into the app for the participant to complete
  Arms: Device

SUMMARY:
The purpose of this study is to compare the short-term changes in gait parameters and functional outcomes after total knee arthroplasty between those who use the StepRite device and those who follow a standard therapy program without the device.

DETAILED DESCRIPTION:
Total Knee Arthroplasty (TKA) is a procedure commonly used in severe degeneration of the knee joint due to osteoarthritis. With an increasing number of TKA's performed in a population that is aging during a time where the amount of healthcare dollars allotted to rehabilitation is declining, there is a need to develop remote monitoring of rehabilitation and to engage and optimize self-management of recovery.

Current management of TKA recovery is typically performed in the out-patient setting and is highly protocol driven. A typical case might be seen by the physical therapist 2-3x/week for 8-10 weeks to perform specific exercises and to monitor progress (i.e. compliance with range of motion (ROM) and strengthening exercises). One recent study suggested that variation in patients' independent exercise and activity after arthroplasty surgery may contribute to variable functional gains.

Telerehabilitation is an emerging method of delivering healthcare. It is likely to become more prevalent as technology improves and funding for clinic appointments diminishes. Recent studies have shown that telerehabilitation can be as effective as conventional treatment, as is well tolerated by both patients and healthcare professionals.

The StepRite system developed by MedHab (http://www.medhab.com/) allows the physical therapist to monitor physical activity and exercise remotely, thereby reducing the need for frequent out-patient visits. A thin insole placed inside the shoe measures foot contact pressure and a small device attached to the shoe measures acceleration. This information is translated into quantitative feedback about exercise compliance and performance measures comparing the surgical side with the non-surgical side. Real time feedback during exercise and weight-bearing activities is provided to the patient, and a HIPAA secured user interface website also displays this information in an online dashboard for both physical therapists and the physician.

Given the potential for improving patient engagement with rehabilitation, this study proposes a treatment model which includes monitoring activity outside of the clinic using the StepRite device and using a combination of outpatient appointments and remote consultations with therapists.

Hypothesis

Patients who use the device post-surgery will demonstrate superior short-term improvements (i.e. 6 months post TKA) with respect to self-reported functional outcomes and gait parameters, compared to a control group who does not use the device.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral total knee arthroplasty performed under regional (spinal +/- epidural) or general anesthesia. Surgical approach via an anterior 4-6 inch incision and utilizing a medial parapatellar arthrotomy incision. Posterior stabilized total knee arthroplasty decision.
* Age 55-75 yr. old
* BMI <35

Exclusion Criteria:

* History of neuromuscular disorder (e.g. Parkinson's, Polio, or stroke).
* Contralateral degenerative joint disease requiring a TKA.
* Pregnancy

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Powers, PhD, Principal Investigator — University of Southern California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device | Usual and Customary Care
Started | 1 | 3
Completed | 0 | 0
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Study terminated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device | Usual and Customary Care | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Knee Osteoarthritis Outcome Score (KOOS)
Description: The KOOS is a validated tool to measure pain and quality of life in patients after TKA
Time Frame: Baseline, 4, 10, 24 weeks
Population: Due to early termination, no evaluable data was collected
Arm/Group | Device | Usual and Customary Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Device | Usual and Customary Care
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3

LIMITATIONS AND CAVEATS:
Early termination lead to no final outcome measures being collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No